CLINICAL TRIAL: NCT06997874
Title: Clinical- and Cost-effectiveness, Safety and Acceptability of Sequential Vitrectomy and Cataract Surgery vs Combined Phacovitrectomy for Rhegmatogenous Retinal Detachment: Randomised Equivalence Trial
Brief Title: Treatment of Retinal Detachment in People Who Have Not Had Cataract Surgery With Vitrectomy vs Vitrectomy and Cataract Removal
Acronym: COMBAT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Northern Ireland Clinical Trials Unit (Other)
Responsible Party: Principal Investigator, Noemi Lois, Clinical Professor of Ophthalmology, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B25/03; ISRCTN13728688 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2025-05-08; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: Rhegmatogenous retinal detachment; phacovitrectomy; vitrectomy; cataract; vitreoretinal surgery
MeSH Terms: conditions — Cataract | interventions — Vitrectomy

STUDY DESIGN:
Intervention Model Description: Pragmatic randomised equivalence trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phacovitrectomy (Active Comparator)
  Interventions: Procedure: Phacovitrectomy
- Vitrectomy (Active Comparator)
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Phacovitrectomy — Participants will undergo phacovitrectomy to remove the lens (phacoemulsification and intraocular lens implantation) and to repair the RRD (vitrectomy). Although a phacovitrectomy is done in the same manner whether the condition to be treated is macular hole or RRD, the calculations required for the surgeon to select which intraocular lens should be implanted are different if there is a RRD with a detached macula. For this reason, a Standard Operating Procedure (SOP) will be prepared for the phacovitrectomy group to guide surgeons on how to best determine the intraocular lens under these circumstances (17). Vitrectomy with any gauge size (e.g.23g, 25g, 27g) will be allowed for the surgery, as per standard care at the participating site. The choice of the tamponade agent will be at the discretion of the treating vitreoretinal surgeon, as per standard care.
  Arms: Phacovitrectomy
Procedure: Vitrectomy — Participants will receive vitrectomy to repair their RRD. The vitrectomy would be done as per standard care. Vitrectomy with any gauge size (e.g.23g, 25g, 27g) will be allowed for the surgery, as per standard care at the participating site. The choice of the tamponade agent will be at the discretion of the treating vitreoretinal surgeon, as per standard care. Then, if a cataract develops, phacoemulsification and intraocular lens implantation will be done as per standard clinical practice.
  Arms: Vitrectomy

SUMMARY:
Background and study aims The retina is the layer at the back of the eye that allows us to see. Sometimes, it can detach from the wall of the eye, causing a condition called rhegmatogenous retinal detachment (RRD), which leads to vision loss and requires surgery. The most common surgery for RRD is vitrectomy, but this can lead to complications like cataracts, which worsen over time and need to be removed with another surgery. Cataract surgery involves replacing the cloudy lens with a clear artificial one. Currently, it's unclear whether it's better to perform both surgeries at the same time or separately. The COMBAT study aims to find out which approach is best by comparing the outcomes of patients who have vitrectomy alone versus those who have both surgeries (vitrectomy and cataract surgery by phacoemulsification and intraocular lens [IOL] implantation) together.

Who can participate? Adults aged 50 and older who have RRD but are not highly myopic (less than -6 diopters or an axial length of 26.5 mm or less) and have not had previous vitreoretinal surgery. Participants must be scheduled for a pars plana vitrectomy to repair their RRD.

What does the study involve? Participants will be randomly assigned to one of two groups: one group will have vitrectomy first and, if needed, cataract surgery later; the other group will have both surgeries at the same time. The study will compare their vision, the number of successful retina reattachments, health related and visual related quality of life, patient satisfaction, complications, additional surgeries and procedures, and costs.

DETAILED DESCRIPTION:
Background Rhegmatogenous retinal detachment (RRD) is the separation of the retina from the wall of the eye, where it is normally attached. It affects 10-18 people per 100,000 per year. Thus, in the UK, with a population of around 68 million, there are 6700-12,000 RRD per year.

RRD can lead to permanent central and peripheral vision loss (i.e. total blindness) if not treated in a timely manner. Vitrectomy is the most common surgery done for RRD. Retinal reattachment following one vitrectomy occurs in 80-88% of eyes, with 59-67% gaining vision above 0.3 LogMAR, which is the vision required to fulfil UK driving standards.

Data from the British and Eire Association of Vitreo-Retinal Surgeons (BEAVRS) showed that most patients with RRD are phakic: they still have their natural lens (i.e. have not had cataract surgery). Data from the BEAVRS database (unpublished, but accessible to the COMBAT research group) showed that of 8436 vitrectomies done in non-high myopic phakic eyes out of 13,900 vitrectomies performed at several sites in the UK, only 10% combined vitrectomy with cataract surgery (called phacovitrectomy) at the time of the RRD repair. Of 664 phakic eyes with at least 12 months follow-up in which combined surgery was not performed at the time of RRD surgery, 320 (48%) were recorded to have a cataract or to have had it already removed within three months of the original vitrectomy. Only 20% of these eyes had their own clear natural lens at 12 months following vitrectomy. Therefore, phacovitrectomy is done in a minority of patients at the time of RRD repair; and many patients have either a cataract present or undergo separate cataract surgery soon after the RRD surgery.

Previous studies have shown the potential benefits of doing combined RRD and cataract surgery. If the cataract is removed when the RRD is repaired, the view of the back of the eye may be clearer, because the surgeon will see through the clear artificial lens. The purpose of the vitrectomy is to remove the vitreous, which is a gel-like structure that fills the back of the eye. The vitreous is involved in the occurrence of the RRD and, given that the vitreous is also present around the posterior part of the lens of the eye, removing the lens allows a more thorough removal of the vitreous. This has the potential to improve the anatomical outcome of the vitrectomy (i.e. reattachment of the retina) and reduce the number of surgeries required because there would be less need for reoperations (repeated vitrectomies) if the first vitrectomy fails to put the retina back in place. Phacovitrectomy would also obviate the need to do the cataract surgery at a later time following the vitrectomy. Adding a phaco to the vitrectomy will add approximately 8 minutes to the surgical time but could save 6000 cataract surgeries per year to the NHS. Moreover, when cataract surgery is done after vitrectomy, the vitreous is no longer present and there is less support to the lens. This may make the cataract surgery more difficult and increase the risk of intraoperative complications.

However, some studies have suggested that postoperative inflammation, accumulation of fluid in the centre of the retina (cystoid macular oedema), epiretinal membrane formation, and posterior synechiae (adherence of the iris to the intraocular lens) may be more frequent after phacovitrectomy. Calculation of the required artificial intraocular lens, which is used to replace the natural lens of the eye during cataract surgery, may be less accurate when doing combined phacovitrectomy in eyes where the macula (i.e. the central retina) is detached. This is because the calculation of the intraocular lens requires measuring the length of the eye and this is less accurate if the macula is detached. However, errors appear to depend on the technique used for this calculation. A less accurate measure of the intraocular lens would mean people may need glasses to improve their vision following surgery.

Rationale for the Study Previous studies comparing vitrectomy with phacovitrectomy in people with RRD have been mostly retrospective and small, with methodological weaknesses. None have addressed patient reported outcomes, patient views and acceptability for one surgery over the other, or costs.

Two systematic reviews of phacovitrectomy versus vitrectomy and subsequent cataract surgery have been published recently. Farahvash et al. included studies in which vitrectomy or phacovitrectomy were used for a variety of retinal disorders, including RRD, macular hole, epiretinal membrane, and others. They included six retrospective before and after studies and one prospective study on RRD but no randomised trials. Results for the RRD group were not given separately. The Mirshahi et al. review included studies specifically comparing surgeries in people with RRD. The review included five retrospective before and after studies, one study defined as a "quasi randomised" and one randomised trial. Only one of the studies included in the review by Mirshahi et al. was in the Farahvash et al. review. The randomised trial in Mirshahi et al. review was a small poorly reported study with 59 patients (59 eyes) randomised to vitrectomy alone (n=29) or phacovitrectomy (n=30). Although not clearly stated, the trial seems to have been a non-inferiority trial with a non-inferiority margin of 10% or less between groups for the primary outcome (retinal reattachment with a single surgery at 6 months). However, a 10% difference in single surgery success on retinal re-attachment seems clinically important. The authors stated that, accepting a 5% type 1 error and 80% power, a sample size of 50 eyes would be needed to detect differences between groups in the primary outcome. Secondary outcomes included final best-corrected visual acuity (BCVA), intraocular pressure, central macular thickness, and progression of cataract in the vitrectomy only group. Mora et al. stated that all outcomes (primary and secondary) were assessed at 1 week and 1, 3 and 6 months after surgery. The trial found no differences in outcomes at six months postsurgery except progression of cataract in the vitrectomy group. Patient reported outcomes and patient experience and acceptability, intra and post-operative complications and costs were not systematically evaluated.

Authors of both systematic reviews called for randomised trials to determine the best surgical approach for people with phakic RRD. COMBAT is such a trial.

Rationale for the Intervention Phacovitrectomy (i.e. phaco to remove the cataract and insert an intraocular lens and vitrectomy to repair the retinal detachment) is performed routinely throughout the UK to treat people with a idiopathic macular hole. However, it is not the standard procedure for people with phakic, non-highly myopic RRD.

Rationale for the Comparator Current standard care in the UK is vitrectomy without concomitant cataract extraction), as shown by data from the BEAVRS database.

Research Hypothesis Combined phacovitrectomy will be preferred by patients because it will provide faster visual recovery and obviate the need for a second surgery (the cataract surgery) following RRD repair, and possibly reduce the number of reoperations related to failure to re-attach the retina. Phacovitrectomy may also reduce other health inequalities because if cataract surgery is required after RRD repair, long waiting times for this surgery in the NHS could adversely affect people with lower income who may be unable to achieve visual rehabilitation as quickly as those with higher income who can afford to have their cataracts removed privately.

Research Question In people with non-highly myopic phakic RRD (Population) in whom vitrectomy is planned to repair their RRD, is phacovitrectomy (Intervention) equivalent (equivalence margin +/- 7 ETDRS letters) to vitrectomy and subsequent cataract surgery (phacoemulsification) if/when needed (Comparator) for improving vision following surgery (primary Outcome) but superior for other outcomes in the 52 weeks (+/- 6 weeks) after surgery.

Study aim To conduct a pragmatic randomised trial evaluating clinical and cost-effectiveness, safety and acceptability and patient experience of combined phacovitrectomy vs vitrectomy and subsequent cataract surgery (if/when needed) for non-highly myopic phakic RRD and to undertake a structured analysis of strategies to implement the phacovitrectomy pathway, if this is shown to be as good or better than current standard care.

Study Objectives In people presenting with a phakic, non-highly myopic RRD, the objectives of the COMBAT study are To determine if the clinical effectiveness of phacovitrectomy is equivalent (or superior) to vitrectomy and subsequent cataract surgery (if/when needed).

To compare the cost-effectiveness of phacovitrectomy vs vitrectomy and subsequent cataract surgery (if/when needed).

To evaluate the participant experience and acceptability of phacovitrectomy compared with vitrectomy and subsequent cataract surgery (if/when needed).

To evaluate the post-trial implementation and scalability of phacovitrectomy.

Study Design Pragmatic, allocation-concealed, single-masked (outcome assessors), multicentre, randomised, equivalence trial with an internal pilot to assess feasibility of recruitment.

Internal Pilot The internal pilot will take place during the first nine months of recruitment, to assess feasibility of recruitment and determine if the study should continue to a full trial. The progression criteria will be assessed nine months after the first site is open to recruitment. The target recruitment will be an average of 0.5 participants per month per open site. With staggered opening of sites, the recruitment target for the pilot is 63 participants (23% of the required sample size for the full trial). Criteria for progression to the full trial are GREEN (Average recruitment rate/site/month: 0.5; number of sites opened: 24; number of participants recruited: 63): Progress to full trial.

AMBER (0.25-0.49; 12-23; 31-62): Discuss feasibility with the TSC and NIHR and develop a recovery plan to reach the recruitment target, including evaluating options to improve recruitment and considering number of eligible patients identified, percentage of these patients randomised and reasons for non-randomisation, site recruitment performance, and recruitment procedures.

RED (<0.25; <12; <31): Decision to progress will be made by the TSC and NIHR.

Study Setting Recruitment for COMBAT will take place in at least 30 hospital eye services (HES) across the four UK nations, with catchment areas that cover diverse populations.

Sequence Generation When a potentially eligible person with a RRD is identified, they will be informed about COMBAT. If they are willing to take part, informed consent will be obtained, and eligibility confirmed. If eligible, the baseline visit will be undertaken (as soon as possible and before the surgery) and participants will be randomised (1:1) to receive phacovitrectomy or vitrectomy. An automated system with the allocation concealed to the ophthalmologist recruiting the participant will be used to generate the random allocation sequence. Minimisation will be used to balance allocation across treatment groups for potentially important factors including centre, surgeon's experience (consultant/vitreoretinal fellow), presenting BCVA (BCVA ≥ 69 ETDRS letters [Snellen equivalent ≥ 20/40; logMAR ≥ 0.3], 24-68 ETDRS letters [Snellen equivalent ≤20/50-20/320; logMAR 0.4-1.2], <24 ETDRS letters [Snellen equivalent <20/320]); macular status (macula on & fovea on, macula off & fovea on, fovea off <7 days, fovea off 7-14 days, fovea off 15-30 days, fovea off >30 days); and presence/absence of PVR-C.

Allocation Concealment An automated system will be used to generate the random allocation sequence. This will conceal the allocation from the ophthalmologist.

Allocation Implementation Each participant will be allocated their own unique trial identifier during the randomisation process, which will be used throughout the study for participant identification on all data collection forms and questionnaires. The patient's allocation will be provided only to unmasked staff (e.g. the surgeon, theatre team).

Definition of Study Eye The unit of randomisation will be the participant, not the eye. In participants with RRD in both eyes, if both eyes are eligible, the "study eye" will be the eye with the best BCVA. If both eyes have the same BCVA, the study eye will be, arbitrarily, the right eye. If both eyes are eligible, the fellow eye would be treated, if possible, in the same way as the study eye. This would apply also if the fellow eye does not have a RRD at presentation but develops it during the trial period (i.e. the participant will be offered the same type of surgery in the fellow eye to that received in the Study Eye, provided that this is pertinent and the participant agrees).

Recruitment Strategy COMBAT will include at least 30 sites. Considering that urgent vitreoretinal cases and specifically RRD are currently done by vitreoretinal fellows in the UK, vitreoretinal fellows will be allowed to take part in the trial. Potentially eligible participants will be identified by members of the direct care team from urgent optometry referrals, from Eye Casualty and from Retina and Vitreoretinal clinics at participating sites. A member of the COMBAT team will then meet with potential participants who express interest in taking part in COMBAT to provide verbal and written details about the trial, including the Participant Information Leaflet (PIL). An audio version of the PIL will be made available where required. If a participant is eligible and provides informed consent, they will be enrolled in the trial. As part of the consent process, patients will be asked if they agree to be invited, at a later date, to take part in a series of 3 (maximum) interviews. Participants will also be asked if, following completion of their participation in the COMBAT trial, data collected as part of their standard care, can be used for future follow-up research.

Screening Procedure All screening data will be recorded via electronic data capture (EDC) to document all participants screened for the study and all participants recruited. Participants screened and not recruited to the study will be documented via EDC, including reasons for not being enrolled. A minimal dataset will be recorded for non-recruited patients, including Age, Sex at Birth, Sexual Orientation, Ethnicity, Preferred language, Socioeconomic Status (e.g. Employment Status, Education level) and partial post code (with the exception of those in Scotland) to determine if there are differences with those willing to participate and recruited. Consent will not be requested to collect this full minimal dataset as data is fully anonymised and is partially collected as part of standard care. Where these data are not routinely collected, participants will be provided with a brief questionnaire and consent will be implied by its completion and return.

Informed Consent COMBAT will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki. Eligible participants may only be included in the trial after written informed consent is obtained. Informed consent must be obtained prior to conducting any trial specific interventions.

Process Evaluation with the Purpose of Informing Implementation A process evaluation focused on the provider perspective of phacovitrectomy will be carried out to assess how the treatment pathways were delivered, barriers and facilitators to implementation, and the influence of local service and wider contexts in implementing phacovitrectomy.

Firstly, semi-structured, theory-driven interviews will be carried out with multidisciplinary groups of healthcare providers, including surgeons, nurses and service managers. These will start 6-12 months after a site starts recruitment to COMBAT, allowing them to develop a level of familiarisation with the service. At the start of recruitment to the trial, these staff will be asked to record important items they needed to put in place at their site to allow implementation of trial procedures (e.g. training of staff to carry out biometry on people with macula-off RRD). Data collection will be guided by the updated Consolidated Framework for Implementation Research (CFIR), which allows systematic study of barriers and drivers to intervention implementation. Secondly, a structured analysis of the required skills and resources and wider strategies used to introduce phacovitrectomy and support implementation over time will be carried out by a study researcher using the ERIC framework (Expert Recommendations for Implementing Change). Together with analysis of barriers and facilitators, and patient data about treatment experience and acceptability; this will assist the development of an implementation blueprint for phacovitrectomy, which would be ready if the COMBAT results favour phacovitrectomy. It is likely to include strategies related to training staff to carry out biometry on people with macula-off RRD and to influence the attitude of surgeons towards phacovitrectomy for non-highly myopic, phakic, RRD.

Sample Size COMBAT is powered to demonstrate treatment equivalence for the primary outcome. Based on two one-sided t-tests at the 2.5% significance level, a 15.2-letter standard deviation and an equivalence margin of +/- 7 ETDRS letters (with a difference of 7 or fewer letters being considered not clinically meaningful), 248 participants would be required to be 90% sure that the 95% confidence interval will exclude a difference in means of more than 7 ETDRS letters. Allowing for 10% dropout, this requires at least 276 participants. This will be sufficient to detect a difference of 16% in the rate of retinal reattachment surgery between groups, which is clinically relevant.

Studies Within a Trial (SWATs) Cochrane reviews of recruitment and retention for randomised trials found little evidence for strategies targeting underserved groups and what limited evidence is available is methodologically poor. Greater inclusion of underserved populations is also a NIHR Equality, Diversity and Inclusion (EDI) strategic priority and meeting this need will require evidence of the effects of strategies that might be used. One observational ("SWAT A") and one intervention SWAT ("SWAT B) will be included in COMBAT to target recruitment and retention of underserved groups. SWAT A will record the proportion in each of the demographic groups who are recruited and retained at each site. Rewards will be offered to the best performing site teams over the recruitment period. Information will be collected on how often the translated PIL are used and whether people for whom these are used are recruited and retained. SWAT B will evaluate whether an EDI-informed PIL increases the recruitment of underserved groups compared to the standard PIL. COMBAT sites that are willing to take part in this SWAT will be asked to use the modified or the standard PIL, in a random order generated by the study statistician. Detailed procedures for the SWATs will be recorded outside of the study protocol and made publicly available with a statistical analysis plan before analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥50 years of age
* Non-highly myopic (< -6 diopters; ≤26.5 mm axial length) phakic RRD
* Naive to previous vitreoretinal surgery
* Pars plana vitrectomy is planned to repair their RRD

Exclusion Criteria:

* Presence of a "formed/established cataract." A "formed/established cataract" is defined as a cataract that, based on the Age-Related Eye Disease Study (AREDS) Research Group, is graded as nuclear sclerosis of >3 and/or if there is an anterior cortical cataract and/or a subcapsular posterior cataract involving the visual axis.
* Pseudophakia or aphakia
* High myopia (≥ -6 diopters; >26.5 mm axial length)
* Giant retinal tear (i.e. presence of one or more retinal tears of >3 clock hours in size)
* Retinal dialysis
* Inclusion in an investigational drug study
* Declined consent for participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2028-05-08 (Estimated); Study Completion 2028-05-08 (Estimated)

PRIMARY OUTCOMES:
Best-Corrected Visual Acuity (BCVA) | 52 weeks (+/- 6 weeks) after surgery
  Change in Best-Corrected Visual Acuity (BCVA) in the affected study eye from baseline to 52 weeks (+/- 6 weeks) after surgery (equivalence margin +/- 7 ETDRS letters)

SECONDARY OUTCOMES:
Primary anatomical success | 52 weeks (+/- 6 weeks) after surgery
  Proportion of eyes with an attached retina after one vitrectomy
Final anatomical success | 52 weeks (+/- 6 weeks) after surgery
  Proportion of eyes with an attached retina after two or more vitrectomies
Intraoperative complications | By 52 weeks (+/- 6 weeks) after surgery
  Total number and by severity score
Postoperative complications | By 52 weeks (+/- 6 weeks) after surgery
  Total number and by severity score
Surgery | By 52 weeks (+/- 6 weeks) after surgery
  Number and type of surgeries performed
Refractive error | 12 weeks after surgery in the phaco-vitrectomy arm and 6-8 weeks post-cataract surgery, if this takes place, as per standard of care, in the vitrectomy only arm
  Difference between aimed (sought) and obtained post-operative refraction
BCVA <69 letters | 52 weeks (+/- 6 weeks) after surgery
  Proportion of participants with BCVA <69 letters
BCVA <34 letters | 52 weeks (+/- 6 weeks) after surgery
  Proportion of participants with BCVA <34 letters
'Best vision' | By 52 weeks (+/- 6 weeks) after surgery
  Time to achieve 'best vision'
BCVA from baseline over time | By 52 weeks (+/- 6 weeks) after surgery
  Change in BCVA from baseline over time
Health related quality of life | 52 weeks (+/- 6 weeks) after surgery
  Measured using EuroQol-5 level (EQ-5D-5L)
Vision-specific quality of life | 52 weeks (+/- 6 weeks) after surgery
  Measured using the National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25)
Participant's experience and acceptability of treatments (including use of Theoretical Framework of Acceptability Questionnaire) | Seriel interviews at week 6, 12 and 52 post-surgery and TFA questionnaire at week 52 post-surgery.
  A mixed methods evaluation of participant experience and treatment acceptability will include serial semi-structured interviews, conducted with a selection of participants. The interview schedule will cover i. Experiences of treatment over time, and factors influencing these experiences ii. Treatment characteristics, consequences and outcomes that are important to participants, and how these vary over time iii. Perceptions about the impact of treatment on their quality of life, including influences on physical, social, and emotional functioning, relationships, employment, civic and recreational activities iv. Acceptability of treatments (informed by Sekhon's framework) including perceptions of effectiveness, burden, affective attitude to the treatment, coherence/understanding of the treatment, and self-efficacy v. Treatment preferences
  The interview data will inform the adaptation of the generic Theoretical Framework of Acceptability (TFA) questionnaire.
Use of health and social care services (including using the MODRUM measure) | From baseline to 52 weeks (+/- 6 weeks) after surgery
  The ModRUM will be used to measure a participant's use of healthcare relating to their eyes. The ModRUM is a validated, concise, generic, measure designed to collect self-report data on the healthcare services people use in UK-based studies Questionnaires will be self-completed by participants with large font questionnaires used when required.
  Worksheets developed for COMBAT will be used to record healthcare use, including for example, surgery costs, ophthalmology, optometrist and other outpatient visits, and GP and nurse consultations.
  Unit costs from publicly available sources will be used (e.g. NHS Reference Costs), for health and social care and will be inflated to current prices where necessary and presented in £ sterling.
Non-healthcare costs to the participants (using a study specific Patient Cost Questionnaire) | To be completed by patients at 12 weeks and 52 weeks after surgery.
  A study specific Patient Cost Questionnaire will be developed to collect non-healthcare costs to the participant. This will measure the out-of-pocket costs to the participant when they attend hospital appointments relating to their eyes and the impact on their ability to work or undertake usual activities. Questionnaires will be self-completed by participants with large font questionnaires used when required.
Safety (of surgery) | By 52 weeks (+/- 6 weeks) after surgery
  Intraoperative and postoperative complications of cataract surgery and vitrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Noemi Lois, Principal Investigator — Wellcome-Wolfson Institute for Experimental Medicine, Queen's University Belfast, Belfast, UK
Locations (27):
- United Kingdom (27):
  - Buckinghamshire Healthcare NHS Trust, Aylesbury
  - Belfast Health and Social Care Trust, Belfast
  - Sandwell and West Birmingham Hospitals NHS Trust, Birmingham
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - County Durham and Darlington NHS Foundation Trust, Darlington
  - NHS Greater Glasgow & Clyde, Glasgow
  - Hull University Teaching Hospitals NHS Trust, Hull
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals Leicester NHS Trust, Leicester
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust, London
  - Guys & St Thomas NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Royal Berkshire NHS Foundation Trust, Reading
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - South Tyneside and Sunderland NHS Trust, Sunderland
  - Mid & South Essex NHS Foundation Trust, Westcliff-on-Sea
  - The Royal Wolverhampton NHS Trust, Wolverhampton
  - York and Scarborough Teaching Hospitals NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: Yes
Following publication of the primary and secondary outcomes and after data has been fully exploited by the COMBAT research team, there may be scope to conduct additional analyses on the data collected. In such instances, formal requests for data will need to be made in writing to the Chief Investigator via the NICTU. If there are requests for data sharing, these will be reviewed on a case-by-case basis by the CI and NICTU (Northern Ireland Clinical Trials Unit, 7 Lennoxvale, Belfast, UK) with approval by the Sponsor required before data are shared.
Access Criteria: Following publication of the primary and secondary outcomes and after data has been fully exploited by the COMBAT research team, there may be scope to conduct additional analyses on the data collected. In such instances, formal requests for data will need to be made in writing to the Chief Investigator via the NICTU. If there are requests for data sharing, these will be reviewed on a case-by-case basis by the CI and NICTU (Northern Ireland Clinical Trials Unit, 7 Lennoxvale, Belfast, UK) with approval by the Sponsor required before data are shared.

REFERENCES:
- See also: COMBAT trial — https://nictu.hscni.net/service/combat/
- Available data/document: Study Protocol: COMBAT trial — https://nictu.hscni.net/service/combat/